CLINICAL TRIAL: NCT01920776
Title: Focused Ultrasound in Septic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, XIiaoting Wang, Dr, Peking Union Medical College Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LHMBCSDXJS-SEPTIC SHOCK
Record Dates: First submitted 2013-08-01; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Septic Shock
Keywords: critical ultrasound
MeSH Terms: conditions — Shock, Septic

ARMS (1):
- Rutine treatment group, Ultrasound group (Experimental)
  Interventions: Other: ultrasound examination; Other: Ultrasound group

INTERVENTIONS:
Other: ultrasound examination
Other: Ultrasound group — Ultrasound group will receive ultrasound examination at least once a day, the results will be noted to the attending who is in charge of the treatment.

SUMMARY:
The investigators hypothesize that lung ultrasound and echocardiography will benefit the septic shock patients by making the treatment more precisely and rapidly. Septic shock patients from multicenter will be enrolled in the study. They will be randomly divided into two groups. The routine treatment group will receive routine treatment according to the SSC guideline. The study group will receive additional ultrasound examination, which will decide the improvement of therapy. Therapy change based on ultrasound results and the prognosis will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* age>18yr
* survive more than 24hrs
* fulfilled septic shock

Exclusion Criteria:

* age < 18yr
* pregnant
* DNR

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
mortality | 28day

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital ICU, Beijing, China

REFERENCES:
- [Derived] Du W, Wang XT, Long Y, Liu DW. Efficacy and Safety of Esmolol in Treatment of Patients with Septic Shock. Chin Med J (Engl). 2016 Jul 20;129(14):1658-65. doi: 10.4103/0366-6999.185856. PMID 27411452